CLINICAL TRIAL: NCT00884026
Title: Pulse Wave Analysis and Augmentation Index Changes Associated With Neuraxial Anesthesia in the Parturient
Brief Title: Can Augmentation Index (AIx) be Used to Predict Hypotension After Spinal Anesthesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H08-03019
Record Dates: First submitted 2009-04-03; First posted 2009-04-20 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hypotension; Cesarean Delivery
Keywords: Cesarean delivery; hypotension; Augmentation Index; Pulse Wave analysis; spinal anesthesia; Hypotension following spinal anesthesia for cesarean delivery
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects that experience hypotension after spinal anesthesia.
  Interventions: Device: AIx measurement with a Sphygmacor TM
- 2 (Active Comparator): Subjects that do not experience hypotension after spinal anesthesia.
  Interventions: Device: AIx measurement with a Sphygmacor TM

INTERVENTIONS:
Device: AIx measurement with a Sphygmacor TM — All subjects will have their AIx measured prior to surgery. After 30 subjects are recruited, they will be split into 2 groups. Group 1 will be those subjects who developed hypotension, and Group 2 will be those subjects who did not develop hypotension. We will then look at the preoperative measured AIx to determine whether there is a baseline difference between the two groups. A threshold value of the AIx with the best sensitivity and specificity for prediction of hypotension will then be determined.
  Arms: 1
Device: AIx measurement with a Sphygmacor TM — The second part of the study will then use the threshold AIx value found from the subjects who developed hypotension from the first 30 subjects to prospectively predict hypotension after spinal anesthesia in another 60 subjects
  Arms: 2

SUMMARY:
A fall in blood pressure (hypotension) occurs in one third of spinal anesthetics administered to pregnant patients undergoing cesarean delivery. However, predicting which patients will experience hypotension following spinal anesthesia has proven difficult. Pulse wave analysis is a repeatable and reproducible method for investigation of cardiovascular function. A device called a SphygmacorTM can be used to measure pulse. The pulse measurement is called the Augmentation Index (AIx). AIx has been useful in detecting risks associated with blood pressure changes after complex surgery in patients with heart and blood vessel disease. In this study the investigators wish to see if it is possible to predict if a subject will experience hypotension based on her AIx measurement preoperatively.

DETAILED DESCRIPTION:
At BC Women's Hospital (BCWH), anesthesiologists give spinal anesthesia for most elective cesarean deliveries. When the spinal medication is given, blood vessels expand in reaction to the spinal medication causing blood pressure to fall. If a patient experiences this common reaction, the anesthesiologist would administer some medications to restore blood pressure to normal. They do this to protect the blood supply to the placenta and to the baby.

It is not known why this happens in some people and not in others. The way blood circulates through the body can provide information about changes occurring in the body. Pulse measurements are a simple way of providing physicians with important clinical information about patient health.

A device called a SphygmacorTM can be used to measure a pulse. The pulse measurement is called the Augmentation Index (AIx). AIx has been useful in detecting risks associated with blood pressure changes after complex surgery in patients with heart and blood vessel disease. In our study we wish to see if AIx can predict a normal patient's risk of hypotension after spinal anesthesia. If a trend between AIx and the onset of hypotension after spinal anesthesia can be found, anesthesiologists can more effectively prevent and treat hypotension by being able to predict whether it will occur.

Consenting subjects will have their blood pressure and AIx measurement taken prior to surgery.

Surgery will commence as per usual practice at BCWH. If hypotension occurs after the spinal anesthesia, anesthesiologist will treat as per usual practice.

Following recruitment and data collection on the first 30 subjects we will review their anesthetic records to assess whether they became hypotensive or not (systolic BP > 20% from baseline). This will give us two groups. Group 1 will be those subjects who developed hypotension, and Group 2 will be those subjects who did not develop hypotension. We will then look at the preoperative measured AIx to determine whether there is a baseline difference between the two groups. A threshold value of the AIx with the best sensitivity and specificity for prediction of hypotension will then be determined.

The second part of the study will then use the threshold AIx value found from the subjects who developed hypotension from the first 30 subjects to prospectively predict hypotension after spinal anesthesia in another 60 subjects.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing elective or urgent cesarean delivery under spinal anesthesia
* Singleton Pregnancy
* Greater than 37 weeks gestation
* Healthy subjects with ASA 1 & 2 classification of health
* Potential subjects need to be able to read and understand English unless independent (non-partner) translator available

Exclusion Criteria:

* ASA 3 or above
* Emergency cesarean delivery for fetal heart rate abnormalities
* Cesarean delivery under general, epidural, or combined spinal epidural anesthesia
* Maternal age <19 years
* Maternal infection
* Mothers with vascular disease - including hypertension/pre-eclampsia
* Mothers with Diabetes Mellitus
* Polyhdramnios
* Multiple Pregnancy
* Height < 150cm or > 180cm
* BMI > 40

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of hypotension following spinal anesthesia. Defined as systolic BP > 20% from baseline. | 1 week

SECONDARY OUTCOMES:
Augmentation Index as measured by the SphygmacorTM preoperatively; Bradycardia requiring pharmacological treatment; Ephedrine requirement; Phenylephrine requirement; Block Height; Nausea/vomiting | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD, FRCPC, Principal Investigator — University of British Columbia; James Shannon, FCARSCI MSc, Study Director — University of British Columbia; Joanne Douglas, MD, FRCPC, Study Director — University of British Columbia; Jessica Tyler, BSc, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital Dept of Anesthesia, Vancouver, British Columbia, Canada